CLINICAL TRIAL: NCT00014365
Title: The Food-Effect Bioavailability Study of Ro 31-7453, a Novel Cell Cycle Inhibitor, in Stable Patient Volunteers With Solid Tumors
Brief Title: Ro 31-7453 in Treating Patients With Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 00-118; CDR0000068537 (Registry Identifier: PDQ (Physician Data Query)); ROCHE-NP15980C; NCI-G01-1928
Record Dates: First submitted 2001-04-10; First posted 2004-04-29 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

INTERVENTIONS:
Drug: MKC-1

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Randomized phase I trial to determine if Ro 31-7453 is more effective with or without food in treating patients who have metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the impact of food on the bioavailability of Ro 31-7453 in patients with locally advanced or metastatic solid tumors.

OUTLINE: This is a randomized, crossover study. Patients are randomized to one of two treatment arms. Arm I: Patients receive oral Ro 31-7453 under fasting conditions on day 1. After a 1-week washout period, patients receive oral Ro 31-7453 under fed conditions. Arm II: Patients receive fed treatment as in arm I on day 1. After a 1-week washout period, patients receive fasted treatment as in arm I. Both arms: At the start of week 3, patients may continue to receive oral Ro 31-7453 every 12 hours on days 1-4. Treatment repeats every 3 weeks for at least 24 weeks in the absence of disease progression or unacceptable toxicity. Patients are followed at 7 days.

PROJECTED ACCRUAL: A total of 10 patients (5 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed locally advanced or metastatic solid tumor for which no standard therapy is available No CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Hemoglobin at least 9 g/dL WBC at least 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) AST and ALT no greater than 1.5 times ULN (4 times ULN for liver metastases) Alkaline phosphatase no greater than 2.5 times ULN (4 times ULN for liver or bone metastases) Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No history or clinical signs of significant cardiovascular disease Other: No other serious concurrent illness No greater than grade II neuropathy No evidence of gastrointestinal dysfunction No intolerance to a high-fat meal Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 3 weeks since prior biologic therapy Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas) Endocrine therapy: At least 2 weeks since prior endocrine therapy (except for antiandrogen therapy) Concurrent antiandrogen therapy allowed Concurrent corticosteroids allowed if stable dose for at least 2 weeks prior to study Radiotherapy: At least 3 weeks since prior radiotherapy Surgery: Not specified Other: No prior enrollment in this study At least 4 weeks since prior investigational drugs No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-10; Primary Completion 2001-10 (Actual); Study Completion 2001-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Soignet, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States